CLINICAL TRIAL: NCT05230030
Title: IMPROV-ing The Impostor Phenomenon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 30194
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-06

CONDITIONS: Impostor Phenomenon
Keywords: Medical trainee; Wellness; Resilience; Burnout; Stress; Physician wellness; Medical education; Observational cohort
MeSH Terms: conditions — imposter syndrome; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Two-part study, starting with observational cohort measuring baseline parameters longitudinally. The second part of the study includes intervention in a single-arm among participants who completed baseline parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational (No Intervention)
- Improvisation Workshops (Experimental): Participants will take part in an improvisation curriculum containing a uniquely designed series of flexibly-timed improvisation workshops administered during the study period. Using published guidelines, workshops will have groups of approximately 10 study participants and last on average 2 hours under the instruction of an expert medical improvisation facilitator.
  Interventions: Behavioral: Improvisation Workshop

INTERVENTIONS:
Behavioral: Improvisation Workshop — Each improvisation workshop will involve a series of exercises derived from an improvisation game book previously developed by study investigators, followed by a reflective debrief of the experience.
  Arms: Improvisation Workshops

SUMMARY:
The impostor phenomenon refers to feelings of self-doubt and fraudulence in one's own abilities, despite the presence of external evidence to suggest otherwise. Symptoms of the impostor phenomenon can impede achievement of career-related goals in medical trainees and impact resilience, stress levels, and burnout. If these symptoms go unnoticed, they could progress to a severity that threatens sustained wellness among medical trainees. Our research questions are: 1) Is the time of the academic year (e.g., beginning, middle, end) associated with severity in impostor phenomenon as measured by the Clance Impostor Phenomenon Scale (CIPS) in medical trainees at the University of Toronto? 2) Is participation in improvisation workshops over the course of an academic year a feasible intervention to mitigate symptoms of impostor phenomenon in medical trainees at the University of Toronto? Combined, our two-part study will explore peak risk periods of impostor phenomenon and whether improvisation workshops are a feasible intervention to address this.

DETAILED DESCRIPTION:
Part 1 of the study:

This will be a prospective cohort study investigating the longitudinal prevalence and levels of impostor phenomenon among medical trainees over the course of one calendar year. Outcomes of interest will be measured in each participant every 3 months with rolling recruitment into the study until the end of the study. Recruitment will last for 2 years. Study investigators will offer and administer an electronic survey to measure impostor phenomenon and symptoms using validated scales. The surveys will be administered to all consenting medical trainees participating in University of Toronto-affiliated hospital rotations on the first day of the rotation. Participant recruitment will occur at University of Toronto-affiliated medical school and hospitals.

Part 2 of the study:

Among participants invited for research question 1 of our study, 10-20 participants will be recruited to further explore the feasibility of an improvisation curriculum during medical training. If volunteer numbers exceed 20, participants will be randomly chosen from the group of interested participants. This curriculum will be a uniquely designed series of flexibly-timed improvisation workshops administered during the study period. Based on within-study participant feedback, sessions will be organized to develop optimal timing and duration of improvisation sessions. Previous studies on improvisation in medical education have varied in terms of timing, frequency, and exercises. Accordingly, each improvisation workshop will involve a series of exercises derived from an improvisation game book previously developed by study investigators, followed by a reflective debrief of the experience. Although improvisation workshops can vary as described, a recently published scoping review revealed three consistent structural elements that will serve as a framework for the improvisation intervention in this study: orientation and setup, culture of safety, and debriefing. Pre-session readings will orient participants to key principles and skills in improvisation. During the exercises, facilitators foster a culture of safety by normalizing uncertainty, creating a low-stakes environment, and providing freedom for time-outs. Improvisation exercises will be followed by debrief to reflect on the session, exchange feedback, and draw connections between improvisation and the impostor phenomenon.

The workshops for this study are designed based on the recommendations established by previous studies with improvisation in medical education. Using published guidelines, workshops will have groups of approximately 10 study participants and last on average 2 hours under the instruction of an expert medical improvisation facilitator. Improvisation sessions will be initially planned to be delivered once per month for 2 hours for four consecutive months with built-in flexibility with respect to session duration and frequency based on participant feedback. Additional sessions can be subsequently offered biweekly and/or for longer than 4 months (up to 10 months) as needed.

ELIGIBILITY:
Inclusion Criteria:

* Have official registration with the University of Toronto Undergraduate or Postgraduate Medical Education offices

Exclusion Criteria:

* Non-fulltime student status
* Exclusion criteria will include participating in the "Improv(ing) the Impostor Phenomenon" study as a co-investigator or concurrent participation in a structured unrelated improvisation program, workshop series, or class outside of the study (ex. The Second City Training Programs/Classes)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Impostor phenomenon score | 3 months
  Score measured by the Clance Impostor Phenomenon Scale; scores can range from 20-100, with higher scores indicating more intense symptoms of impostor phenomenon

SECONDARY OUTCOMES:
Resilience score | 3 months
  Score measured by the Connor-Davidson Resilience Scale; scores can range from 0-100, with higher scores meaning higher resilience
Perceived stress score | 3 months
  Score measured by the Perceived Stress Scale; scores can range from 0-40, with higher scores meaning higher perceived stress
Burnout | 3 months
  Measured by the Maslach Burnout Inventory-Human Services Survey -2 for Medical Personnel with no quantitative score

CONTACTS AND LOCATIONS:
Overall Officials: Esther Bui, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mullangi S, Jagsi R. Imposter Syndrome: Treat the Cause, Not the Symptom. JAMA. 2019 Aug 6;322(5):403-404. doi: 10.1001/jama.2019.9788. No abstract available. PMID 31386138
- [Background] LaDonna KA, Ginsburg S, Watling C. "Rising to the Level of Your Incompetence": What Physicians' Self-Assessment of Their Performance Reveals About the Imposter Syndrome in Medicine. Acad Med. 2018 May;93(5):763-768. doi: 10.1097/ACM.0000000000002046. PMID 29116983
- [Background] Gottlieb M. More than meets the eye: The impact of imposter syndrome on feedback receptivity. Med Educ. 2021 Feb;55(2):144-145. doi: 10.1111/medu.14412. Epub 2020 Nov 18. No abstract available. PMID 33155297
- [Background] Gottlieb M, Chung A, Battaglioli N, Sebok-Syer SS, Kalantari A. Impostor syndrome among physicians and physicians in training: A scoping review. Med Educ. 2020 Feb;54(2):116-124. doi: 10.1111/medu.13956. Epub 2019 Nov 6. PMID 31692028
- [Background] Clance PR, Imes SA. The imposter phenomenon in high achieving women: Dynamics and therapeutic intervention. Psychotherapy: Theory, Research & Practice. 1978;15(3):241. doi:10.1037/h0086006
- [Background] Clance P. The Impostor Phenomenon: Overcoming The Fear That Haunts Your Success. Atlanta, Ga.: Peachtree Publishers; 1985.
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Maslach C, Jackson S, Leiter M. Maslach Burnout Inven- tory Manual. 3rd ed. Palo Alto: Consulting Psychologists Press; 1996.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417